CLINICAL TRIAL: NCT00436852
Title: A Phase II Study of ABT-751, an Orally Bioavailable Tubulin Binding Agent, in Children With Relapsed or Refractory Neuroblastoma
Brief Title: ABT-751 in Treating Children With Neuroblastoma That Has Relapsed or Not Responded to Previous Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANBL0621; NCI-2009-00402 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI-07-C-0074; CDR0000529858 (Other: Clinical Trials.gov); NCI-P6554; U10CA098543 (NIH); COG-ANBL0621 (Other: Children's Oncology Group)
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Results first posted 2014-02-28 (Estimated); Last update posted 2019-07-17 (Actual); Status verified 2019-07

CONDITIONS: Disseminated Neuroblastoma; Recurrent Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — ABT751; E 7010

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Measurable disease by CT or MRI scan (ABT-751 chemotherapy) (Experimental): Patients receive oral ABT-751 (200 mg/m2) once daily on days 1-7. Treatment repeats every 21 days for 52 courses in the absence of disease progression or unacceptable toxicity. Quality-of-life assessment at baseline and prior to each course of treatment. A pharmacological study (pharmacokinetic profile of ABT-751) will be determined.
  Interventions: Drug: ABT-751; Procedure: quality-of-life assessment
- Evaluable by I-MIBG scintigraphy (ABT-751) (Experimental): Patients receive oral ABT-751 (200 mg/m2) once daily on days 1-7. Treatment repeats every 21 days for 52 courses in the absence of disease progression or unacceptable toxicity. Quality-of-life assessment at baseline and prior to each course of treatment. A pharmacological study (pharmacokinetic profile of ABT-751) will be determined.
  Interventions: Drug: ABT-751; Procedure: quality-of-life assessment

INTERVENTIONS:
Drug: ABT-751 — Given orally
  Other Names: E7010
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This phase II trial is studying how well ABT-751 works in treating children with neuroblastoma that has relapsed or not responded to previous treatment. Drugs used in chemotherapy, such as ABT-751, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the time to disease progression in children with refractory or relapsed neuroblastoma treated with ABT-751 vs historical controls.

SECONDARY OBJECTIVES:

I. Determine the objective response rate in patients with measurable disease treatment with this drug.

II. Determine whether ABT-751 improves quality of life of these patients. III. Determine the toxicity of ABT-751. IV. Determine the pharmacokinetic profile of ABT-751 in these patients.

OUTLINE:

Patients receive oral ABT-751 once daily on days 1-7. Treatment repeats every 21 days for 52 courses in the absence of disease progression or unacceptable toxicity.

Blood is collected periodically during course 1 for pharmacokinetic studies. Quality of life is assessed at baseline and prior to each course of treatment.

After completion of study treatment, patients are followed up for up to 5.1 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed neuroblastoma meeting the following criteria:

  * Refractory or relapsed disease
  * No curative treatment option and no additional therapy proven to prolong survival with an acceptable quality of life is available
  * Evidence of disease progression (enlargement of existing measurable tumors or the appearance of new tumors) during prior treatment OR biopsy-proven viable neuroblastoma if stable disease but refractory to prior treatment
* Previously irradiated soft tissue or bony lesion must meet ≥ 1 of the following criteria:

  * Viable neuroblastoma determined by biopsy ≥ 6 weeks after radiation therapy
  * Growth in the lesion determined by CT scan or MRI
* Measurable or evaluable disease

  * Measurable disease is defined as ≥ 20 mm in ≥ 1 dimension by MRI, CT scan, or x-ray OR ≥ 10 mm in ≥ 1 dimension by spiral CT scan
  * Evaluable disease is defined as iodine I 123 metaiodobenzylguanidine (^123I MIBG)-positive lesion at ≥ 1 site

    * Must not have measurable disease by CT scan or MRI
  * No elevated urinary catecholamines and/or bone marrow evidence of tumor, without measurable or evaluable disease by imaging modalities (CT scan, MRI, or ^123I MIBG)
* Karnofsky performance status (PS) 50-100% (> 16 years of age) OR Lansky PS 50-100% (≤ 16 years of age)
* Life expectancy ≥ 8 weeks
* Hemoglobin ≥ 7.5 g/dL (transfusions allowed)
* Absolute neutrophil count > 250/mm³
* Platelet count > 25,000/mm³ (without platelet transfusion support for ≥ 7 days)
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT < 5 times ULN
* Creatinine normal for age and gender as follows: OR creatinine clearance or radioisotope glomerular filtration rate ≥ 60 mL/min

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months-11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male])
* Shortening fraction ≥ 27% by echocardiogram
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective double-barrier contraception during and for 90 days after completion of study treatment
* Seizure disorder allowed if controlled and receiving anticonvulsants
* Neurologic toxicity from prior therapy or tumor involvement ≤ grade 2
* No evidence of active graft-vs-host disease
* No allergy to sulfa-containing medications
* No known HIV positivity
* No clinically significant unrelated systemic illness (e.g., serious infection) that would limit study compliance
* Concurrent filgrastim (G-CSF) allowed if medically indicated
* Recovered from all prior therapy
* No prior ABT-751
* More than 2 weeks since prior myelosuppressive chemotherapy
* More than 7 days since prior anticancer biologic agents (e.g., retinoids)
* More than 4 weeks since prior palliative radiation therapy (small port) or therapeutic ^123I MIBG
* More than 6 weeks since prior substantial radiation therapy (> 50% pelvis, craniospinal, or total-body radiation)
* More than 4 months since prior allogeneic stem cell transplantation (SCT) (2 months for autologous SCT) and recovered

  * Infusion of autologous peripheral blood mononuclear cells without high-dose chemotherapy or preparative regimen is not considered SCT
* More than 30 days since prior investigational drug therapy
* More than 30 days since prior immunotherapy (monoclonal antibody therapy or vaccine therapy)
* More than 1 week since prior growth factor treatment
* No other concurrent anticancer agents, including chemotherapy, immunomodulating agents, or biologic therapy (retinoids)
* No concurrent radiation therapy, including palliative radiation therapy
* No concurrent treatment for graft-vs-host disease
* No concurrent epoetin alfa, sargramostim (GM-CSF), or interleukin-11

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 92 (Actual)
Dates: Start 2007-01; Primary Completion 2010-09-01 (Actual); Study Completion 2015-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Fox, MD, Principal Investigator — Children's Oncology Group
Locations (12):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - C S Mott Children's Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Cook Children's Medical Center, Fort Worth, Texas
- Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Disease Evaluable by I-MIBG Scintigraphy (ABT-751); Measurable Disease by CT or MRI Scan (ABT-751): Patients receive oral ABT-751 (200 mg/m2) once daily on days 1-7. Treatment repeats every 21 days for 52 courses in the absence of disease progression or unacceptable toxicity. Quality-of-life assessment at baseline and prior to each course of treatment. A pharmacological study (pharmacokinetic profile of ABT-751) will be determined.
Period: Overall Study
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Started | 45 | 47
Completed | 10 | 2
Not Completed | 35 | 45
Not completed — Death | 23 | 34
Not completed — Lack of Efficacy | 9 | 7
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: The protocol-specified definition of evaluability was applied. This was not an intention-to-treat analysis because patients who did not receive study drug were excluded (inevaluable).
Groups:
- Total: Total of all reporting groups
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751) | Total
Number analyzed (Participants) | 45 | 47 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 42 | 45 | 87
  Between 18 and 65 years | 3 | 2 | 5
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 8.46 [6.23 to 12.91] | 7.55 [5.91 to 12.43] | 8.00 [6.07 to 12.67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 21 | 35
  Male | 31 | 26 | 57
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 35 | 41 | 76
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 9 | 17
  White | 30 | 30 | 60
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  United States | 45 | 36 | 81
  Canada | 0 | 10 | 10
  Jamaica | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression as Assessed by Response Evaluation Criteria in Solid Tumors
Description: Median time to progression observed on ABT-751, along with 95% confidence intervals.
Time Frame: From time to enrollment to death due to any cause, assessed up to 5.1 years
Population: as for baseline characteristics
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Disease Evaluable by I-MIBG Scintigraphy (ABT-751); Measurable Disease by CT or MRI Scan (ABT-751): Patients who met study eligibility criteria and receive at least one dose of oral ABT-751 were evaluable for the efficacy analysis.
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Number analyzed (Participants) | 44 | 47
days | 45 [42 to 85] | 42 [36 to 56]

2. Primary Outcome: 1-year Progression-free Survival
Description: PFS probabilities calculated using the Kaplan-Meier method, along 95% confidence intervals, separately for each stratum.
Time Frame: From the day of enrollment to the date of disease progression/recurrence , or the date of death (all causes of mortality) if disease progression/recurrence is not reached, assessed up to 1 yr. Pts were to be followed for 5 yrs after completion of therapy
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Number analyzed (Participants) | 44 | 47
percent probability | 19 [7 to 31] | 7 [0 to 15]

3. Secondary Outcome: Objective Response Rate
Description: The percentage of patients who are responders will be tabulated, including a 95% confidence interval on the percentage. Responders were defined as patients who achieved a best overall response of complete response (CR) or partial response (PR) at any time on the study including patients who achieved ≥PR and later had progressive disease or relapse. Response in patients with measurable disease will be assessed by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0 or by Curie criteria for measuring response by MIBG scans in patients with evaluable disease by 123I-MIBG scan. Per RECIST: CR= Disappearance of all target lesions; PR= at least 30% decrease in the sum of the longest diameter of target lesions. Per Curie criteria: CR= complete resolution of all MIBG positive lesions; PR= resolution of at least one MIBG positive lesion with persistence of other MIBG positive lesions.
Time Frame: Duration of protocol therapy, up to 3 years
Population: Patients who met study eligibility criteria and received at least one dose of oral ABT-751 were evaluable for the response analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of patients
Groups:
- Disease Evaluable by I-MIBG Scintigraphy (ABT-751): Patients with evaluable disease by (123)I-MIBG scintigraphy (positive at a minimum of one site) with or without bone marrow metastases but without RECIST (Response Evaluation in Solid Tumors) measureable disease.
- Measurable Disease by CT or MRI Scan (ABT-751): Patients with RECIST measurable disease on CT or MRI scan, with or without (123)I-MIBG positive disease, with or without bone marrow metastases.
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Number analyzed (Participants) | 43 | 47
Percentage of patients | 12 [2 to 21] | 2 [0 to 6]

4. Secondary Outcome: Quality of Life Measured by PedsQL™ Generic Core Scale Version 4.0
Description: The QOL score will be reverse linearly transformed to a 0-100 percentage point scale (0=100, 1=75, 2=50, 3=25, 4=0), with higher scores indicating better health-related quality of life, and the average of all 23 items will be calculated as the composite score.
Time Frame: At baseline
Population: Eligible patients with a QOL evaluation at baseline were included in the analysis.
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Number analyzed (Participants) | 37 | 34
Scores on a scale | 80 [44 to 99] | 68 [29 to 100]

5. Secondary Outcome: Percentage of Participants With Grade 3 or Higher Toxicity
Description: Percentage of patients with at least one Grade 3 or higher toxicity, as assessed by Common Terminology Criteria for Adverse Events version 3.0, will be tabulated.
Time Frame: From enrollment until 30 days after the end of protocol therapy
Population: All eligible patients who received at least 1 dose of ABT-751 were evaluable for toxicity and included in the analysis.
Measure: Number; unit: Percentage of patients
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Number analyzed (Participants) | 44 | 47
Percentage of patients | 75.0 | 72.3

6. Secondary Outcome: Pharmacokinetics of ABT-751: Cmax
Description: Values of the maximum observed concentration (Cmax) will be determined for the first dose.Descriptive statistics for these variables will be provided.
Time Frame: After the first dose of ABT-751, at 0.5, 1, 2, 3, 5, 8, 10-12, and 24 hours post-dose.
Population: All eligible patients from Group 1 (Disease Evaluable by I-MIBG Scintigraphy (ABT-751)) and Group 2 (Measurable Disease by CT or MRI Scan (ABT-751)) who received the first dose of ABT-751 and participated in the pharmacokinetic studies were included in the analysis and are presented as a single Group, as the interest was in both groups combined.
Measure: Median (Full Range); unit: mg/ml
Groups:
- All Eligible Patients: All eligible patients who received the first dose of ABT-751 and participated in the pharmacokinetic studies
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 16
mg/ml | 15.3 [7.3 to 22.4]

7. Secondary Outcome: Pharmacokinetics of ABT-751: Tmax
Description: Values of the time to maximum observed concentration (Tmax) will be determined for the first dose.Descriptive statistics for these variables will be provided.
Time Frame: After the first dose of ABT-751, at 0.5, 1, 2, 3, 5, 8, 10-12, and 24 hours post-dose.
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 16
hours | 1 [1 to 3]

8. Secondary Outcome: Pharmacokinetics of ABT-751: AUC
Description: Values of the area under concentration time curve [AUC(0-∞)] will be determined for the first dose. Descriptive statistics for these variables will be provided.
Time Frame: After the first dose of ABT-751, at 0.5, 1, 2, 3, 5, 8, 10-12, and 24 hours post-dose.
Population: as for outcome 6
Measure: Median (Full Range); unit: mg·hours/ml
Arm/Group | All Eligible Patients
Number analyzed (Participants) | 16
mg·hours/ml | 77.5 [46.8 to 169.3]

ADVERSE EVENTS:
Arm/Group | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) | Measurable Disease by CT or MRI Scan (ABT-751)
Serious Adverse Events (participants affected / at risk) | 3/44 | 4/47
Other Adverse Events (participants affected / at risk) | 17/44 | 24/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) (N=44) | Measurable Disease by CT or MRI Scan (ABT-751) (N=47)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 1 | 0
" Bronchospasm, wheezing" (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Death not associated with CTCAE term - Death NOS (General disorders) | 1 | 0
Death not associated with CTCAE term - Disease progression NOS (General disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Febrile neutropenia (fever, unk. origin,w/o infection,ANC<1x10e9, fever>=38.5C) (Blood and lymphatic system disorders) | 0 | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 1 | 1
Gait/walking: Extremity-lower (gait/walking) (General disorders) | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 1 | 2
Hemorrhage, GI - Rectum (Gastrointestinal disorders) | 1 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypoglycemia: Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia: Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 0 | 2
Hyponatremia: Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection (clinical or microbiological Dx) w/ Gr 3-4 neutrophils, ANC<1.0x10e9 - Blood (Infections and infestations) | 0 | 1
Infection (clinical or microbiological Dx) w/ Gr 3-4 neutrophils, ANC<1.0x10e9 - Paranasal (Infections and infestations) | 1 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Blood (Infections and infestations) | 2 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Bone (osteomyelitis) (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Catheter-related (Infections and infestations) | 1 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 0 | 1
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (cellulitis) (Infections and infestations) | 2 | 0
Infection with normal ANC or Grade 1 or 2 neutrophils - Upper airway NOS (Infections and infestations) | 2 | 0
Infection with unknown ANC - Blood (Infections and infestations) | 0 | 1
Infection with unknown ANC - Middle ear (otitis media) (Infections and infestations) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 1
Left ventricular systolic dysfunction (Cardiac disorders) | 1 | 1
Mood alteration - Agitation (Psychiatric disorders) | 1 | 0
Mood alteration - Anxiety (Psychiatric disorders) | 0 | 1
Mood alteration - Depression (Psychiatric disorders) | 0 | 1
Muscle weakness, generalized or specific area (not due to neuropathy) - Whole body/generalized (Musculoskeletal and connective tissue disorders) | 1 | 0
Neuropathy: sensory (Nervous system disorders) | 1 | 4
Obstruction, GI - Small bowel NOS (Gastrointestinal disorders) | 0 | 2
Pain - Abdomen NOS (Gastrointestinal disorders) | 1 | 0
Pain - Bone (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 3 | 3
Pain - Head/headache (Nervous system disorders) | 0 | 1
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain - Neuralgia/peripheral nerve (Nervous system disorders) | 0 | 3
Personality/behavioral (Psychiatric disorders) | 1 | 0
Platelets (Investigations) | 1 | 0
Syncope (fainting) (Nervous system disorders) | 1 | 0
Taste alteration (dysgeusia) (Nervous system disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2
Weight loss (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Evaluable by I-MIBG Scintigraphy (ABT-751) (N=44) | Measurable Disease by CT or MRI Scan (ABT-751) (N=47)
Constipation (Gastrointestinal disorders) | 8 (8) | 12 (12)
Anorexia (Metabolism and nutrition disorders) | 7 (7) | 9 (9)
"ALT, SGPT (serum glutamic pyruvic transaminase)" (Investigations) | 9 (9) | 14 (14)
"AST: AST, SGOT(serum glutamic oxaloacetic transaminase)" (Investigations) | 7 (7) | 14 (14)
"Albumin, serum-low (hypoalbuminemia)" (Metabolism and nutrition disorders) | 0 (0) | 12 (12)
"Bicarbonate, serum-low" (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
" Cholesterol: Cholesterol, serum-high (hypercholestremia)" (Investigations) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Creatinine (Investigations) | 0 (0) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 8 (8)
" Fatigue (asthenia, lethargy, malaise)" (General disorders) | 13 (13) | 9 (9)
" Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L)" (General disorders) | 6 (6) | 12 (12)
GGT: GGT (gamma-Glutamyl transpeptidase) (Investigations) | 4 (4) | 4 (4)
Hemoglobin (Blood and lymphatic system disorders) | 12 (12) | 24 (24)
" Hemorrhage, pulmonary/upper respiratory - Nose" (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
"Hypercalcemia: Calcium, serum-high (hypercalcemia)" (Metabolism and nutrition disorders) | 0 (0) | 4 (4)
"Hyperglycemia: Glucose, serum-high (hyperglycemia)" (Metabolism and nutrition disorders) | 7 (7) | 12 (12)
"Hypermagnesemia: Magnesium, serum-high (hypermagnesemia)" (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypertension (Vascular disorders) | 0 (0) | 3 (3)
"Hypertriglyceridemia: Triglyceride, serum-high (hypertriglyceridemia)" (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
"Hypocalcemia: Calcium, serum-low (hypocalcemia)" (Metabolism and nutrition disorders) | 0 (0) | 6 (6)
"Hypoglycemia: Glucose, serum-low (hypoglycemia)" (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
"Hypokalemia: Potassium, serum-low (hypokalemia)" (Metabolism and nutrition disorders) | 4 (4) | 11 (11)
"Hypomagnesemia: Magnesium, serum-low (hypomagnesemia)" (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
"Hyponatremia: Sodium, serum-low (hyponatremia)" (Metabolism and nutrition disorders) | 6 (6) | 14 (14)
"Hypophosphatemia: Phosphate, serum-low (hypophosphatemia)" (Metabolism and nutrition disorders) | 0 (0) | 8 (8)
Infection with normal ANC or Grade 1 or 2 neutrophils - Sinus (Infections and infestations) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 6 (6) | 3 (3)
Leukocytes (total WBC) (Investigations) | 17 (17) | 19 (19)
Lymphopenia (Investigations) | 5 (5) | 10 (10)
Mood alteration - Agitation (Psychiatric disorders) | 0 (0) | 3 (3)
Mood alteration - Anxiety (Psychiatric disorders) | 3 (3) | 0 (0)
Mood alteration - Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 13 (13) | 16 (16)
Neuropathy: sensory (Nervous system disorders) | 12 (12) | 10 (10)
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 17 (17) | 14 (14)
Pain - Abdomen NOS (Gastrointestinal disorders) | 9 (9) | 11 (11)
Pain - Back (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 11 (11) | 11 (11)
Pain - Head/headache (Nervous system disorders) | 7 (7) | 9 (9)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Pain - Stomach (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pain - Throat/pharynx/larynx (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Platelets (Investigations) | 13 (13) | 18 (18)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 6 (6) | 11 (11)
Weight loss (Investigations) | 4 (4) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No